CLINICAL TRIAL: NCT02525393
Title: Safety and Efficacy of Non Invasive Transcranial Brain Stimulation in Motor Stroke Rehabilitation
Brief Title: Transcranial Stimulation in Motor Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Federico Dagata, Assistant Professor, University of Turin, Italy
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI 339
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Stroke
Keywords: Rehabilitation; Non Invasive Brain Stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- tDCS+rTMS (Experimental): Stroke patients were treated with an initial two weeks of transcranial direct current stimulation and after six months with two weeks of repetitive transcranial magnetic stimulation.
  Interventions: Device: tDCS; Device: rTMS
- rTMS+tDCS (Experimental): Stroke patients were treated with an initial two weeks of repetitive transcranial magnetic stimulation and after six months with two weeks of transcranial direct current stimulation.
  Interventions: Device: tDCS; Device: rTMS
- Sham stimulation (Sham Comparator): Stroke patients were treated with two weeks of sham transcranial direct current stimulation.
  Interventions: Device: Sham

INTERVENTIONS:
Device: tDCS — Stroke rehabilitation performed with the aid of a transcranial electrical stimulation device.
  Other Names: HDC Stim device Newronica
  Arms: rTMS+tDCS; tDCS+rTMS
Device: rTMS — Stroke rehabilitation performed with the aid of a repetitive transcranial magnetic stimulation device.
  Other Names: PowerMAG 100 MAG&More
  Arms: rTMS+tDCS; tDCS+rTMS
Device: Sham — Stroke sham stimulation performed with the aid of a transcranial electrical stimulation device.
  Other Names: HDC Stim device Newronica
  Arms: Sham stimulation

SUMMARY:
Patients were randomized in 3 groups: two intervent groups and a control group. The first group received two weeks of daily session of repetitive Transcranial Magnetic Stimulation (rTMS, 10 sessions) and, at least 6 months after, two weeks of daily transcranial Direct Current Stimulation (tDCS, 10 sessions); the second group received 10 daily session of tDCS and, after at least 6 months, 10 sessions of rTMS; the control group received 10 daily session of sham tDCS.

Physiatric evaluations (ARAT scale), neuropsychological assessment and ERP (P300) were performed before (1 week) and after (1 week) the end of each treatment. Furthermore, all patients underwent follow-up neuropsychological assessment 6 months after the end of each stimulation period and follow-up physiatric evaluation at 3 and 6 months after the end of each stimulation period.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke (> 6 months from the accident)

Exclusion Criteria:

* general cognitive impairment (Mini Mental State Examination < 25), severe functional disability (Barthel Index < 45),
* psychiatric disorders,
* degenerative neurological disorders,
* epilepsy,
* severe medical conditions,
* having been implanted a drug infusion system, spinal/brain-stimulator, or endovascular coil

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from the baseline ARAT (measures Grasp, Grip, Pinch, Gross Movement) | Baseline; 1 month; 3 months; 6 months; 6 months and 1 week; 7 months; 9 months; 12 months
  Action Research Arm Test (ARAT) measures Grasp, Grip, Pinch, Gross Movement. Baseline is 1 week before first treatment; other time frame: 1 week after first treatment; 3 months after first treatment; 6 months follow-up after first treatment; 1 week before second treatment; 1 week after second treatment; 3 months follow-up after second treatment; 6 months follow-up after second treatment.

SECONDARY OUTCOMES:
P300 (latency) | Baseline; 1 month; 6 months and 1 week; 7 months
  The P300 (P3) wave is an event related potential (ERP) component elicited in the process of decision making.
  Investigators measured the latency of the component 1 week before first treatment; 1 week after first treatment; 1 week before second treatment; 1 week after second treatment.
Cognition (standardized neuropsychological assessment) | Baseline; 1 month; 6 months; 6 months and 1 week; 7 months; 12 months
  The patients were evaluated by means of a standardized neuropsychological assessment consisting of a battery of cognitive tests involving the following domains: verbal short-term memory, visuospatial learning, working memory, verbal learning, attention and frontal executive functions, and general cognitive impairment.
  The assessment was repeated 1 week before first treatment; 1 week after first treatment; 6 months follow-up after first treatment; 1 week before second treatment; 1 week after second treatment; 6 months follow-up after second treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Federico D'Agata, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Italy